CLINICAL TRIAL: NCT05293405
Title: Neuroinflammatory Imaging Using TSPO PET Tracer in Paients With Autoimmune Encephalomyelitis
Brief Title: Neuroinflammatory PET Imaging in Autoimmune Encephalomyelitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: (2021)CER(375)
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Autoimmune Encephalomyelitis
MeSH Terms: conditions — Encephalomyelitis, Autoimmune, Experimental

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Group (Experimental)
  Interventions: Diagnostic Test: 18F-DPA-714 PET
- Healthy Volunteers Group (Sham Comparator)
  Interventions: Diagnostic Test: 18F-DPA-714 PET

INTERVENTIONS:
Diagnostic Test: 18F-DPA-714 PET — TSPO expression are quantitatively analyzed in all brain regions or spinal cord using 18F-DPA-714 PET

SUMMARY:
Autoimmune encephalomyelitis is a heterogeneous group of central nervous system (CNS) autoimmune diseases characterized by the production of anti-neuron-associated autoantibodies which target neuronal surface proteins, synaptic receptors and intracellular antigens. MRI, as a current first-line imaging tool of CNS inflammation, is difficult to diagnose them because the majority of patients have normal MRI images, and only a few may show local signal or structural abnormalities (including inflammation, edema, or atrophy). The 18 kDa translocator protein (TSPO) expression in the CNS is upregulated in response to microglia activation. DPA-714 is high affinity for binding to TSPO, making 18F-labeled DPA-714 (18F-DPA-714) PET a very promising diagnostic imaging tool for neuroinflammation in patients with autoimmune encephalomyelitis.This study aims to explore the value of 18F-DPA-714 PET in the early diagnosis, therapeutic assessment and prognosis in patients with autoimmune encephalomyelitis.

ELIGIBILITY:
Experimental group:

Inclusion criteria:

1. Patients with onset for less than 2 years
2. Serum autoantibody positive
3. cognitive impairment or movement disorder diagnosed by two or more certified specialists.

Exclusion criteria:

1. Patients who do not meet the clinical、laboratory and imaging criteria of immune-related cognitive and movement disorders
2. Medical history of surgery, trauma, stroke, tumor in brain or spine cord
3. Alcoholism or drug dependence (addiction)
4. Patients with pregnancy

Healthy Volunteers group:

Inclusion criteria:

1. able to understand the purpose of clinical research and test plan
2. In the brain and spine cord MR assessment, it is judged as "normal"

Exclusion criteria:

1. Any major mental illness; history of schizophrenia or schizoaffective disorder
2. Any important neurological disease, such as cerebrovascular disease, inflammation or infectious disease, demyelinating disease, neurodegenerative disease, trauma in brain or spine cord
3. History of alcohol or drug abuse/dependence
4. Medical history of cardiac and lung disease, tumors, blood disease, poorly controlled chronic diseases
5. Patients with pregnancy

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-12-13 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
TSPO expression level | Baseline
  quantitatively assessing the level of neuroinflammation in all brain regions or spinal cord
TSPO expression level | 3 months after baseline
  quantitatively assessing the level of neuroinflammation in all brain regions or spinal cord
TSPO expression level | 12 months after baseline
  quantitatively assessing the level of neuroinflammation in all brain regions or spinal cord

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China

REFERENCES:
- [Derived] Meng H, He L, Chunyu H, Zhou Q, Wang J, Qu Q, Hai W, Zhang Y, Li B, Zhang M, Chen S. 18F-DPA714 PET/MRI as a potential imaging tool for detecting possible antibody-negative autoimmune encephalitis: a prospective study. J Neurol. 2024 Dec;271(12):7592-7604. doi: 10.1007/s00415-024-12690-w. Epub 2024 Sep 19. PMID 39294471